CLINICAL TRIAL: NCT04919590
Title: Text Message Quit Vaping Intervention for Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Truth Initiative (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TruthInitiativeQVSTeen
Record Dates: First submitted 2021-06-04; First posted 2021-06-09 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Vaping; Cessation, Tobacco
Keywords: Vaping cessation; Mobile intervention; Adolescents
MeSH Terms: conditions — Vaping; Tobacco Use Cessation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are not explicitly told they are in the control group, although they may deduce their assignment from presence or lack of regular text message intervention.
  Research staff doing data collection will not be aware of the random assignments and all participants will receive the same follow-up assessments regardless of assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- This is Quitting (Experimental): Participants will be enrolled to receive messages from This is Quitting.
  Users receive one age-appropriate message per day tailored to their enrollment date or quit date, which can be set and reset via text message. Those not ready to quit receive 4 weeks of messages focused on building skills and confidence. Users who set a quit date receive messages for a week preceding it and 8 weeks afterward that include encouragement and support, skill- and self-efficacy building exercises, coping strategies, and information about the risks of vaping, benefits of quitting, and cutting down to quit. Keywords COPE, STRESS, SLIP, and MORE provide on-demand support.
  Interventions: Behavioral: This is Quitting
- Assessment only control (Other): After an initial enrollment message, participants will be contacted monthly to assess e-cigarette use. At the end of the study data collection period, they will receive information on how to sign up for This is Quitting if they are interested in the program.
  Interventions: Other: Assessment only control
- Waitlist control (Other): After an initial enrollment message, participants will receive no contact from study staff except for 1-month and 7-month follow-up assessments. At the end of the study data collection period, they will receive information on how to sign up for This is Quitting if they are interested in the program.
  Interventions: Other: Waitlist control

INTERVENTIONS:
Behavioral: This is Quitting — Text message-based intervention for quit vaping support.
  Arms: This is Quitting
Other: Assessment only control — Assessment only
  Arms: Assessment only control
Other: Waitlist control — No contact until follow-up survey, waitlisted to receive intervention post study
  Arms: Waitlist control

SUMMARY:
This research study, conducted by Truth Initiative, will help us learn how text messaging can help adolescents between 13 and 17 years of age quit vaping.

DETAILED DESCRIPTION:
The Teen Quit Vaping Study (QVS Teen) is a comparative effectiveness trial to evaluate the effectiveness of a quit vaping text message program in promoting abstinence from e-cigarettes among young users aged 13-17. This study is a 3-arm randomized controlled trial conducted among young users aged 13-17 recruited through online channels. Participants will be randomized to a quit vaping text message intervention, an assessment-only control condition, or a waitlist control condition. The primary aim is to examine 30-day point prevalence abstinence at 7-months post enrollment (roughly corresponds to 6-months post-treatment).

ELIGIBILITY:
Inclusion Criteria:

* Age 13-17
* Past 30-day use of e-cigarettes containing nicotine
* Interest in quitting e-cigarette use in the next 30 days
* US residence

Exclusion Criteria:

* Failure to confirm mobile number after initial sign-up

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1681 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Truth Initiative, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
IPD are not available to other researchers. For access to deidentified dataset, please contact study administrator for more information.

REFERENCES:
- [Background] Graham AL, Cha S, Jacobs MA, Amato MS, Funsten AL, Edwards G, Papandonatos GD. A Vaping Cessation Text Message Program for Adolescent E-Cigarette Users: A Randomized Clinical Trial. JAMA. 2024 Sep 3;332(9):713-721. doi: 10.1001/jama.2024.11057. PMID 39110436
- [Derived] Graham AL, Cha S, Do EK, Jacobs MA, Edwards G, Papandonatos GD. Dual abstinence from nicotine vaping and cannabis use among young people: secondary analyses from two U.S.-based randomized controlled trials of vaping cessation. Subst Abuse Treat Prev Policy. 2025 Nov 3;20(1):48. doi: 10.1186/s13011-025-00679-1. PMID 41177894

RESULTS

PARTICIPANT FLOW:
Groups:
- This is Quitting: Participants will be enrolled to receive messages from This is Quitting.
  Users receive one age-appropriate message per day tailored to their enrollment date or quit date, which can be set and reset via text message. Those not ready to quit receive 4 weeks of messages focused on building skills and confidence. Users who set a quit date receive messages for a week preceding it and 8 weeks afterward that include encouragement and support, skill- and self-efficacy building exercises, coping strategies, and information about the risks of vaping, benefits of quitting, and cutting down to quit. Keywords COPE, STRESS, SLIP, and MORE provide on-demand support.
  This is Quitting: Text message-based intervention for quit vaping support.
Period: Overall Study
Arm/Group | This is Quitting | Assessment Only Control | Waitlist Control
Started | 759 | 744 | 178
Completed | 759 | 744 | 178
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Waitlist Control: After an initial enrollment message, participants will be contacted only for data collection at 1 and 7 months post enrollment. At the end of the study data collection period, they will receive information on how to sign up for This is Quitting if they are interested in the program.
  Waitlist only
- Total: Total of all reporting groups
Arm/Group | This is Quitting | Assessment Only Control | Waitlist Control | Total
Number analyzed (Participants) | 759 | 744 | 178 | 1681
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 759 | 744 | 178 | 1681
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.4 (0.8) | 16.4 (0.8) | 16.4 (0.8) | 16.4 (0.8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 386 | 369 | 93 | 848
  Gender: Male | 314 | 314 | 69 | 697
  Gender: Non-binary or Other | 51 | 59 | 16 | 126
  Gender: Unknown or not reported | 8 | 2 | 0 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 11 | 7 | 3 | 21
  Asian | 16 | 20 | 4 | 40
  Native Hawaiian or Other Pacific Islander | 3 | 2 | 1 | 6
  Black or African American | 76 | 76 | 15 | 167
  White | 469 | 461 | 117 | 1047
  More than one race | 139 | 136 | 26 | 301
  Unknown or Not Reported | 45 | 42 | 12 | 99
Region of Enrollment [Number; unit: participants]
  United States | 759 | 744 | 178 | 1681

OUTCOME MEASURES:

1. Primary Outcome: Self-reported 30-day Point Prevalence Abstinence
Description: In the past 30 days, did you vape at all, even a puff of someone else's?
Time Frame: 7 months post enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | This is Quitting | Assessment Only Control | Waitlist Control
Number analyzed (Participants) | 759 | 744 | 178
Participants | 287 | 208 | 49

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | This is Quitting | Assessment Only Control | Waitlist Control
All-Cause Mortality (participants affected / at risk) | 0/759 | 0/744 | 0/178
Serious Adverse Events (participants affected / at risk) | 0/759 | 0/744 | 0/178
Other Adverse Events (participants affected / at risk) | 0/759 | 0/744 | 0/178

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-07): https://cdn.clinicaltrials.gov/large-docs/90/NCT04919590/Prot_SAP_000.pdf